CLINICAL TRIAL: NCT05579899
Title: A Randomized, Vehicle-controlled, Safety and Efficacy Study of EVO101 in Adult Subjects With Atopic Dermatitis
Brief Title: Safety and Efficacy Study of EVO101 Topical Cream in Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evommune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVO101-AD001
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Matching vehicle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EVO101 Cream (Experimental): Active Treatment, BID, 8 weeks
  Interventions: Drug: EVO101
- Vehicle Cream (Placebo Comparator): Vehicle Treatment, BID, 8 weeks
  Interventions: Drug: EVO101

INTERVENTIONS:
Drug: EVO101 — Topical Cream

SUMMARY:
This is a Phase 2a safety and efficacy study of EVO101 for the treatment of adults with atopic dermatitis

DETAILED DESCRIPTION:
This is a Phase 2a safety and efficacy study of EVO101 Topical Cream, 0.1%, applied twice daily for 8 weeks in adults with mild-to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant, non-lactating females, age 18 years or older
2. Chronic atopic dermatitis for at least 1 year
3. IGA score of 2 or 3
4. BSA of AD involvement of 4-12%
5. EASI of 5-20

Exclusion Criteria:

1. Significant AD flare with 4 weeks
2. Use of biologic therapy within 12 weeks
3. Regular use of tanning booth within 4 weeks
4. Skin condition that could interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Bauer, MD, Study Director — Evommune, Inc.
Locations (21):
- United States (21):
  - Saguaro Dermatology, Phoenix, Arizona
  - Clinical Trials Institute of Northwest Arkansas, Fayetteville, Arkansas
  - Northwest AR Clinical Trials Center, PLLC, Rogers, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Metropolis Dermatology, Los Angeles, California
  - Dermatology Research Associate, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research, LLC, Coral Gables, Florida
  - Lenus Research and Medical Group, Miami, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - SkinSpecialists, LLC, Omaha, Nebraska
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - Dermatologists of Southwest Ohio, Mason, Ohio
  - Oregon Medical Research Center, Portland, Oregon
  - DermResearch, Austin, Texas
  - J&S Studies, Inc, College Station, Texas
  - Center for Clinical Studies, Ltd LLC, Houston, Texas
  - Pariser Dermatology Specialists, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Following publication
Access Criteria: to be determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EVO101 Cream | Vehicle Cream
Started | 60 | 59
Completed | 57 | 51
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVO101 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 55 | 106
  >=65 years | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 23 | 22 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 24 | 44
  Not Hispanic or Latino | 39 | 32 | 71
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Eczema Area and Severity Index (EASI) From Baseline to Week 8
Description: EASI assesses the extent and severity of atopic dermatitis. EASI is a composite index with scores ranging from 0 to 72. Higher values indicate more severe or extensive disease.
Time Frame: 8 weeks
Population: All participants assigned to EVO101 or Vehicle treatment.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | EVO101 Cream | Vehicle Cream
Number analyzed (Participants) | 60 | 59
Percent change from baseline | -43.5 (60.85) | -62.0 (38.78)

2. Secondary Outcome: Investigator Global Assessment (IGA) Response (Number of Participants With >= 2 Points Change From Baseline to Week 8)
Description: The IGA assesses the overall appearance and severity of atopic dermatitis using a 5-point scale [0 (clear) to 4 (severe)]. The outcome measures is reported as the number of participants achieving a reduction of 2 or greater on the IGA from baseline to Week 8.
Time Frame: 8 weeks
Population: Participants assigned to EVO101 or Vehicle with available data at Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | EVO101 Cream | Vehicle Cream
Number analyzed (Participants) | 57 | 51
Participants
  Yes | 20 | 23
  No | 37 | 28

3. Secondary Outcome: Percent Body Surface Area (BSA) Affected by Atopic Dermatitis Over Time, Change From Baseline to Week 8
Description: BSA estimates the extent of atopic dermatitis involvement and is expressed as a percentage of total body surface area. The outcome measure describes the mean change from baseline in percent of the body surface area affected by AD.
Time Frame: 8 weeks
Population: Participants assigned to EVO101 or Vehicle with available data at Week 8
Measure: Mean (Standard Deviation); unit: percentage of total body surface area
Arm/Group | EVO101 Cream | Vehicle Cream
Number analyzed (Participants) | 57 | 51
percentage of total body surface area | -2.1 (6.45) | -3.5 (2.99)

4. Secondary Outcome: Pruritus-NRS, Change From Baseline to Week 8
Description: The pruritus-NRS is an 11-point scale used by subjects to rate their worst itch severity over the past 24 hours with 0 indicating "no itch" and 10 indicating "worst itch imaginable".
Time Frame: 8 weeks
Population: Participants assigned to EVO101 or Vehicle with available data at Week 8
Measure: Mean (Standard Deviation); unit: Change in units on a scale
Arm/Group | EVO101 Cream | Vehicle Cream
Number analyzed (Participants) | 47 | 42
Change in units on a scale | -2.5 (2.16) | -3.5 (2.55)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | EVO101 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 19/60 | 30/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVO101 Cream (N=60) | Vehicle Cream (N=58)
Application site pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (14)
Application site erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 10 (11)
Application site oedema (Skin and subcutaneous tissue disorders) | 3 (3) | 11 (12)
Application site pain (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (8)
Application site dryness (Surgical and medical procedures) | 2 (2) | 8 (8)
Application site exfoliation (Skin and subcutaneous tissue disorders) | 3 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon written approval by Evommune, the PI may publicly disclose site results for only (1) non-commercial and (2) internal scientific research and educational purposes

DOCUMENTS (2):
  • Study Protocol (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05579899/Prot_001.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT05579899/SAP_002.pdf